CLINICAL TRIAL: NCT06580769
Title: Effects on Physical Condition and Body Composition of a Physical Exercise Program Implemented Through Immersive Virtual Reality in University Adults: Protocol for a Randomized Controlled Trial
Brief Title: Effects of an Immersive Virtual Reality Program
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autónoma de Chile (Other)
Responsible Party: Principal Investigator, Andrés Godoy Cumillaf, Principal Investigator, Universidad Autónoma de Chile
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UAChileTco
Record Dates: First submitted 2024-08-21; First posted 2024-08-30 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-08

CONDITIONS: Physical Activity; Virtual Reality; Physical Fitness
Keywords: fat; Muscle; strength; cardiorespiratory fitness
MeSH Terms: conditions — Motor Activity; Platelet Glycoprotein IV Deficiency | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental (Experimental): They will develop the physics activity program through immersive virtual reality
  Interventions: Other: Physical activity
- Experimental 2 (Experimental): They will develop a physical activity program through HIIT
  Interventions: Other: Physical activity
- Control (No Intervention): They do not perform physical activity

INTERVENTIONS:
Other: Physical activity — Implementation of a physical activity program, executed through immersive virtual reality
  Arms: Experimental; Experimental 2

SUMMARY:
A tool that could be useful to eliminate the barriers of not practicing physical activity can be immersive virtual reality, which is characterized by being a technique where a person, through the use of a screen mounted on the head, receives images, sounds and tactile sensations of a simulated world.

In the area of physical exercise, evidence places immersive virtual reality as a tool that encourages healthy behaviors and the practice of physical activity, increasing adherence to exercise in the long term. In addition to the fact that performing physical activity by this means generates a high level of enjoyment in the participants, so if the use of this technology generates enjoyment in those who use it and contributes to complying with the recommendations of physical activity, it is logical to think that a physical exercise program executed through immersive virtual reality could contribute to improving parameters related to people's health. Therefore, the objective of this randomized controlled trial is to evaluate the effect of a physical exercise program carried out through immersive virtual reality on health-related variables.

DETAILED DESCRIPTION:
Physical fitness (PF) is a measure that integrates most of the body's functions that are involved during the performance of any physical activity or physical exercise. Although its variation depends largely on genetic components, the physical exercise factor is one of the environmental conditioning factors that most influence its development. Evidence indicates that adequate PF values are considered important for people's health as they are related to better cardiovascular, skeletal, and mental health, which is why PF is considered an important component of a healthy lifestyle.

On the other hand, there is body composition, which is responsible for quantifying, determining relationships and defining the quantitative changes of the different components of the human body. Its study is important to understand the effect of environmental factors such as growth, diet, diseases and physical exercise on the body. Research that has studied the effects of physical activity interventions aimed at improving PF indicates that they lead to improvements in people's body composition, specifically, reductions in fat and increases in muscle mass. This is beneficial for health, since a greater accumulation of fat in regions such as the waist and abdomen increases the risk factor for the development of metabolic diseases and insulin resistance, while adequate muscle mass values are associated with improvements in the metabolism of hepatic, pancreatic, and immune tissue, among others.

Despite ample evidence exposing the health benefits, more than a quarter of adults worldwide are physically inactive. Among the factors that explain this behavior is that the practice of physical exercise is considered boring and difficult, which together with long working hours, keeps people away from the practice, which added to factors such as lack of motivation, family and social support, nearby sports environments and habits of practicing physical activity, generate negative attitudes towards physical activity, which leads to not practicing it. All of the above increases in university students, a complex population, due to the influence of bad healthy habits as a result of the impact of the academic load, the change from school life to university life and all university obligations.

A tool that could be useful to eliminate the barriers described for not practicing physical activity can be immersive virtual reality (IVR), which is characterized by being a technique where a person, through the use of a screen mounted on the head, receives images, sounds and tactile sensations from a simulated world. all through an avatar that allows movements to be shown in a way that is consistent with the subject's body in a first-person perspective, making participants adjust their real actions in response to the observed movements of the avatar, driven by the illusory sensation of having the avatar's body, which generates measurable motor and physiological responses in the real body. In this sense, the RVI allows us to experience situations that, in reality, due to the necessary time or space, would not be possible.

Several studies have analyzed the benefits of IVR in the field of public health, allowing greater effectiveness in the work of repetitive tasks, graphic and acoustic feedback, and adherence to physical therapies. This has been reflected in several studies that describe the effects of programs implemented through IVR in the rehabilitation of patients with cardiovascular accidents, Parkinson's, fibromyalgia and obstructive pulmonary diseases, among others.

Regarding the area of physical exercise, the evidence places it as a tool that encourages healthy behaviors and the practice of physical activity, increasing adherence to exercise in the long term. A recent scoping review established that its use stimulates moderate and vigorous intensity levels, which could contribute to meeting physical activity recommendations, while other studies conclude that practicing physical exercise through IVR causes moderate and vigorous intensity physical activity, which are the ones that bring health benefits. On the other hand, there is information that indicates that performing physical activity through IVR generates a high level of enjoyment in participants, greater calorie burning, greater concentration and the feeling of being able to continue exercising for longer.

Taking into account that the practice of physical exercise in the adult population is low, even more so in the university population, the IVR could be an alternative way to overcome the limitations that prevent the practice of physical exercise in adults. In addition, if the use of this technology generates enjoyment in those who use it and contributes to complying with the recommendations for physical activity, it is logical to think that a physical exercise program executed through IVR could contribute to improving PF and reducing body fat values and increasing muscle mass. However, the available evidence has not found information describing the effects of running exercise programs through IVR on physical fitness, nor the fat and muscle components of body composition. This study will provide useful information for this emerging line of research. It is hypothesized that the physical exercise program carried out through immersive virtual reality will cause improvements in physical condition and body composition in university adults. The objective of this randomized controlled trial is to evaluate the effect on physical fitness and body composition of a physical exercise program performed through immersive virtual reality in university adults.

ELIGIBILITY:
Inclusion Criteria:

* Be a university student
* Present medical consent authorizing the performance of physical activity
* Signing of informed consent

Exclusion Criteria:

* Have a physical or mental impairment that prevents you from engaging in physical activity
* Have a vision impairment that does not allow you to use the immersive virtual reality
* Belong to a special interest group (professional athletes or pregnant women)

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Physical fitness | From registration to the end of the physical activity intervention, it will be a period of 16 weeks.
  Cardiorespiratory fitness will be measured through the 20-meter shuttle run test, and maximum oxygen consumption will be estimated. Lower body muscle strength will be measured through the long jump test. Upper body muscle strength will be measured through manual grip strength (Takei 5401). Speed/agility will be assessed through the 4x10 test.
Body Composition | From registration to the end of the physical activity intervention, it will be a period of 16 weeks.
  Weight will be evaluated through a scale (Seca 222), with the participant barefoot and with the least possible clothing. Size will be obtained with a height gauge (Seca 222), with the participant barefoot, in an upright position, at the end of a normal inspiration. Both measures will be taken in duplicate, using the mean for statistical analyses.
  Body mass index will be determined by dividing weight by height squared. Waist circumference will be determined at the midpoint between the last rib and the iliac crest. The average of two measurements will be used.
  The percentage of adipose and muscle tissue will be calculated by means of tetrapolar electrical bioimpedance (Tanita MC 780U). It will be complemented by the measurement of body perimeters, bone diameters and skin folds, according to the protocol described by the International Society for the Advancement of Kineanthropometry.

CONTACTS AND LOCATIONS:
Overall Officials: Paola Fuentes-Merino, MsC, Principal Investigator — Universidad Autónoma de Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giakoni-Ramirez F, Godoy-Cumillaf A, Espoz-Lazo S, Duclos-Bastias D, Del Val Martin P. Physical Activity in Immersive Virtual Reality: A Scoping Review. Healthcare (Basel). 2023 May 25;11(11):1553. doi: 10.3390/healthcare11111553. PMID 37297694
- [Result] Godoy-Cumillaf A, Fuentes-Merino P, Giakoni-Ramirez F, Duclos-Bastias D, Merellano-Navarro E. Effectiveness of a physical activity intervention on the overweight and obesity of Chilean schoolchildren. Medicine (Baltimore). 2022 Sep 30;101(39):e30908. doi: 10.1097/MD.0000000000030908. PMID 36181063
- [Result] Sousa CV, Hwang J, Cabrera-Perez R, Fernandez A, Misawa A, Newhook K, Lu AS. Active video games in fully immersive virtual reality elicit moderate-to-vigorous physical activity and improve cognitive performance in sedentary college students. J Sport Health Sci. 2022 Mar;11(2):164-171. doi: 10.1016/j.jshs.2021.05.002. Epub 2021 May 16. PMID 34004390
- [Result] Debska M, Polechonski J, Mynarski A, Polechonski P. Enjoyment and Intensity of Physical Activity in Immersive Virtual Reality Performed on Innovative Training Devices in Compliance with Recommendations for Health. Int J Environ Res Public Health. 2019 Sep 30;16(19):3673. doi: 10.3390/ijerph16193673. PMID 31574911
- [Derived] Godoy-Cumillaf A, Fuentes-Merino P, Giakoni-Ramirez F, Munoz-Strale C, de Souza-Lima J, Duclos-Bastias D, Parra-Saldias M, Bruneau-Chavez J, Merellano-Navarro E. Effects of a Walking-Based Physical Activity Intervention on Health Indicators in University Students: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 Dec 10;14:e83983. doi: 10.2196/83983. PMID 41370823